CLINICAL TRIAL: NCT05166031
Title: A Phase III Study to Evaluate the Immunogenicity and Safety of Concomitant Administration of Two Doses of a Novel Oral Polio Type 2 Vaccine and Bivalent Oral Polio Vaccine in Healthy Infants
Brief Title: Evaluation of the Immunogenicity and Safety of Concomitant Administration of Novel Oral Polio Type 2 Vaccine and Bivalent Oral Polio Vaccine
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decided not to conduct it
Sponsor: Fidec Corporation (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: nOPV2-001-ABMG
Record Dates: First submitted 2020-10-26; First posted 2021-12-21 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bOPV dose (Active Comparator): Naïve infants to receive two doses of bOPV at 2 and 3 months of age.
  Interventions: Biological: bOPV and nOPV2
- nOPV2 dose (Active Comparator): Naïve infants to receive two doses of nOPV2 at 2 and 3 months of age.
  Interventions: Biological: bOPV and nOPV2
- bOPV + nOPV2 dose (Experimental): Naïve infants to receive two doses of nOPV2 and bOPV at 2 and 3 months of age.
  Interventions: Biological: bOPV and nOPV2

INTERVENTIONS:
Biological: bOPV and nOPV2 — Approximately 265 subjects will receive 2 doses of bOPV, nOPV2 or bOPV + nOPV2 per arm separated by 28 days between doses.

SUMMARY:
The study will assess and compare the immune response and safety following the co-administration of Novel Oral Polio Type 2 (nOPV2) and bivalent Oral Polio Vaccine (bOPV) in comparison with nOPV2 or bOPV in infants aged 2 months who have never received vaccination against poliomyelitis.

ELIGIBILITY:
Inclusion Criteria:

1. Infants aged 8 weeks (-1, + 2 weeks) with birth weight >2,500 gm.
2. Healthy infants without obvious medical conditions like immunodeficiency diseases, severe congenital malformations, severe neurological diseases or any other disease that require high doses of corticosteroids or immunotherapies that preclude the subject to be in the study as established by the medical history and physical examination.
3. Written informed consent obtained from 1 or 2 parent(s) or legal guardian(s) as per country regulations.

Exclusion Criteria:

1. Infants who have received previous vaccination according to the National Immunization Program (NIP) (i.e. vaccination against poliomyelitis and/or receipt of diphtheria-tetanus-whole cell pertussis-hepatitis B-Haemophilus influenzae type b [DTPw-HB-Hib vaccine]).
2. Infants with anyone under 10 years of age in their household (living in the same house or apartment unit) who does not have complete "age appropriate" vaccination status with respect to poliovirus vaccines at the time of study vaccine administration according to the Dominican Republic NIP.
3. Infants having a member of their household (living in the same house or apartment unit) who is under 6 months of age at the moment of study vaccine administration.
4. Infants having a member of their household (living in the same house or apartment unit) who has received oral polio vaccine (OPV) in the previous 3 months before study vaccine administration.
5. Any confirmed or suspected immunosuppressive or known immunodeficient condition including human immunodeficiency virus infection in the potential participant or any member of the subject's household.
6. Family history of congenital or hereditary immunodeficiency.
7. Major congenital defects or serious uncontrolled chronic illness (neurologic, pulmonary, gastrointestinal, hepatic, renal, or endocrine).
8. Known allergy to any component of the study vaccines or to any antibiotics, that share molecular composition with the nOPV2 vaccines.
9. Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
10. Acute severe febrile illness at day of vaccination deemed by the Investigator to be a contraindication for vaccination (the child can be included at a later time if within age window and all inclusion criteria are met.).
11. Subject who, in the opinion of the Investigator, is unlikely to comply with the protocol or is inappropriate to be included in the study for the safety or the benefit-risk ratio of the subject.

Ages: 7 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-10-18 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate | 2 months
  Assessment and comparison of seroconversion rate to poliovirus types 1, 2 and 3 28 days following co-administration of two doses of nOPV2 and bOPV with two doses of nOPV2 or two doses of bOPV
Incidence of serious adverse reactions (SARs) , important medical reactions (IMRs) and severe solicited adverse reactions (ARs) | 6 months
  Number of serious adverse reactions, important medical reactions and severe solicited adverse reactions following co-administration of nOPV2 and bOPV in comparison with nOPV2 or bOPV

SECONDARY OUTCOMES:
Immunogenicity to poliovirus type 2 | 2 months
  Assessment and comparison of geometric mean neutralizing antibody titers against poliovirus type 2 following administration of nOPV2 with co-administration of nOPV2 and bOPV
Immunogenicity to poliovirus type 2 | 2 months
  Assessment and comparison of seroconversion rate against poliovirus type 2 following administration of nOPV2 with co-administration of nOPV2 and bOPV
Immunogenicity to poliovirus type 2 | 2 months
  Assessment and comparison of seroprotection rate against poliovirus type 2 following administration of nOPV2 with co-administration of nOPV2 and bOPV
Assessment and comparison of immunogenicity to poliovirus type 1 and 3 | 2 months
  Assessment and comparison of the seroprotection rates against poliovirus types 1 and 3 following administration of bOPV with co-administration of nOPV2 and bOPV.
Assessment and comparison of immunogenicity to poliovirus type 1 and 3 | 2 months
  Assessment and comparison of the geometric mean neutralizing against poliovirus types 1 and 3 following administration of bOPV with co-administration of nOPV2 and bOPV.
Assesment of SAEs, IMEs and any AEs | 6 months
  Number, severity and causality of any serious adverse event (SAE), any solicited AE, any unsolicited AE and any important medical events (IME) following co-administration of nOPV2 and bOPV in comparison with nOPV2 or bOPV
Assessment and comparison of viral shedding | 1 month
  Assessment and comparison of viral shedding in stool at fixed time points following administration of nOPV2, bOPV or the co-administration of nOPV2 and bOPV.